CLINICAL TRIAL: NCT07257237
Title: The Effect of Sleep Hygiene Education on Sleep Quality and Blood Pressure in Patients With Essential Hypertension in a Family Practice Center: A Randomized Controlled Trial
Brief Title: Sleep Hygiene Education and Blood Pressure Control in Essential Hypertension in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozturk Gurer Tutu, MD (Other)
Responsible Party: Sponsor-Investigator, Ozturk Gurer Tutu, MD, Family Medicine Specialist, Mustafa Kemal University
Organization: Mustafa Kemal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MKU-SLEEPHTN-2024
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Essential Hypertension; Sleep Quality; Primary Care
Keywords: hypertension; sleep hygiene; sleep quality; primary care; Pittsburgh Sleep Quality Index; blood pressure; family medicine; behavioral intervention; randomized controlled trial
MeSH Terms: conditions — Essential Hypertension; Sleep Initiation and Maintenance Disorders; Hypertension; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: The trial used an open-label design for participants and family physicians. However, nurses who measured blood pressure as an outcome were blinded to group assignments throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep hygiene education (Experimental): Participants in this arm received a 10-15 minute face-to-face sleep hygiene education session delivered by a family physician during the baseline visit. They were given a printed brochure summarising sleep hygiene recommendations and were asked to keep a sleep diary for 8 weeks. The family physician telephoned participants at weeks 2, 4, and 6 to reinforce adherence to sleep hygiene behaviours.
  Interventions: Behavioral: Sleep hygiene education program
- Usual care (No Intervention): Participants in this arm received usual medical care for essential hypertension according to routine practice in the family practice center. No additional sleep hygiene education, sleep diary, or telephone follow-up related to sleep was provided during the 8-week study period.

INTERVENTIONS:
Behavioral: Sleep hygiene education program — Brief structured education on sleep hygiene principles (regular sleep-wake schedule, limiting caffeine and screen exposure before bedtime, creating a quiet and dark sleep environment), delivered face-to-face by a family physician during the baseline visit, supported by a printed brochure and telephone reinforcement at weeks 2, 4, and 6.
  Arms: Sleep hygiene education

SUMMARY:
This randomized controlled trial evaluated the effect of a brief sleep hygiene education program on sleep quality and blood pressure in adults with essential hypertension attending a family practice center in southern Türkiye. Poor sleep quality is common in patients with hypertension and may contribute to inadequate blood pressure control and increased cardiovascular risk.

In this single-centre trial, 138 adult patients with physician-diagnosed essential hypertension were randomly assigned to an intervention group or a control group. The intervention group received a 10-15 minute face-to-face sleep hygiene education session delivered by a family physician, together with a printed brochure summarising key sleep hygiene recommendations. Participants were asked to keep a sleep diary for 8 weeks and were contacted by telephone at weeks 2, 4, and 6 to reinforce the recommendations. The control group received usual medical care for hypertension without additional education or follow-up contacts.

Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI), and office blood pressure was measured at baseline and after 8 weeks in both groups. The primary objective was to determine whether sleep hygiene education improves sleep quality; secondary objectives were to evaluate the effects of the intervention on systolic and diastolic blood pressure compared with usual care.

DETAILED DESCRIPTION:
Hypertensive patients frequently report poor sleep quality, which may adversely affect blood pressure control and increase cardiovascular risk. Although pharmacological treatment is the cornerstone of hypertension management, simple behavioural interventions such as sleep hygiene education may provide additional benefits in primary care. This single-centre, parallel-group, randomized controlled trial was conducted in a family practice center in southern Türkiye to investigate whether a structured sleep hygiene education program could improve sleep quality and blood pressure among adults with essential hypertension.

Eligible participants were men and women aged 30-65 years with physician-diagnosed essential hypertension who were under regular follow-up at the family practice center. Patients with impaired cognitive function, alcohol or substance dependence, pregnancy, recent changes in antihypertensive medication, active infection or malignancy, or diagnosed obstructive sleep apnea were excluded. After obtaining written informed consent and completing baseline assessments, participants were randomized in blocks of four to an intervention or control group.

The intervention consisted of a 10-15 minute face-to-face education session on sleep hygiene principles (such as regular sleep-wake schedule, limiting caffeine and screen exposure before bedtime, creating a quiet and dark sleep environment) delivered by a family physician. Participants received a printed brochure summarising these recommendations and were asked to keep a daily sleep diary for 8 weeks. The family physician telephoned participants in the intervention group at weeks 2, 4, and 6 to answer questions and reinforce adherence to sleep hygiene behaviours. The control group received usual care for hypertension without additional contact related to sleep hygiene. No changes to antihypertensive medication were made as part of the study protocol.

The primary outcome was change in Pittsburgh Sleep Quality Index (PSQI) global score from baseline to 8 weeks. Secondary outcomes were changes in systolic and diastolic office blood pressure over the same period. Blood pressure was measured using an automated oscillometric device following a standardised protocol, and the mean of three readings taken after 5 minutes of rest was recorded. The study was approved by the Hatay Mustafa Kemal University Clinical Research Ethics Committee, and all participants provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30-65 years
* Physician-diagnosed essential hypertension (office blood pressure >140/90 mmHg or on antihypertensive treatment)
* Under regular follow-up at the family practice center
* At least high school education
* Able and willing to provide written informed consent

Exclusion Criteria:

* Impaired mental capacity or cognitive impairment
* Alcohol or substance dependence
* Pregnancy
* Any change in antihypertensive medication within the previous 2 months
* Active infection or active malignancy
* Diagnosed obstructive sleep apnea

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) global score | From baseline to 8 weeks after randomization
  The Pittsburgh Sleep Quality Index (PSQI) is a self-reported questionnaire assessing sleep quality over the previous month. The global score ranges from 0 to 21, with higher scores indicating poorer sleep quality. The primary outcome is the change in PSQI global score from baseline to 8 weeks in each group and the difference in mean change between groups.

SECONDARY OUTCOMES:
Change in systolic blood pressure (SBP) | From baseline to 8 weeks after randomization
  Office systolic blood pressure (mmHg) measured using an automated oscillometric device following a standardised protocol. Three measurements were taken after 5 minutes of rest, and the mean of the three readings was recorded. The outcome is the change in systolic blood pressure from baseline to 8 weeks and the difference in mean change between groups.
Change in diastolic blood pressure (DBP) | From baseline to 8 weeks after randomization
  Office diastolic blood pressure (mmHg) measured using the same protocol as for systolic blood pressure (three readings after 5 minutes of rest, mean value recorded). The outcome is the change in diastolic blood pressure from baseline to 8 weeks and the difference in mean change between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Dörtyol Özerli Family Health Center, Antakya, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) for all study variables used in the analyses are publicly available in the Zenodo repository. The dataset includes anonymised sociodemographic characteristics, baseline and follow-up PSQI scores, and systolic and diastolic blood pressure measurements for all participants.
Time Frame: The deidentified individual participant data (IPD) and associated data dictionary have been available in the Zenodo repository since 28 July 2025 and will remain publicly accessible for an indefinite period.
Access Criteria: Deidentified IPD and the accompanying data dictionary are openly available to any researcher. Data can be downloaded directly from the Zenodo repository without registration, prior approval, or a data use agreement.
URL: https://doi.org/10.5281/zenodo.16529837

REFERENCES:
- [Derived] Tutu OG, Bilen V, Ozer C. The effect of sleep hygiene education on sleep quality and blood pressure in patients with essential hypertension in a family practice center: a randomized controlled trial. Fam Pract. 2025 Dec 9;43(1):cmaf110. doi: 10.1093/fampra/cmaf110. PMID 41511014
- See also: Zenodo repository: deidentified individual participant data for this trial — https://doi.org/10.5281/zenodo.16529837
- Available data/document: Individual Participant Data Set: 10.5281/zenodo.16529837 — https://doi.org/10.5281/zenodo.16529837 — Deidentified individual participant data set including sociodemographic variables, baseline and 8-week PSQI scores, and systolic and diastolic blood pressure measurements for all randomized participants. Data are shared together with a data dictionary under the license specified on the Zenodo record.